CLINICAL TRIAL: NCT05395429
Title: Clinical Evaluation of Genetron TERT/BRAF PCR Kit in Thyroid Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Genetron Health (Industry)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Yunnan Cancer Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 20210155
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2022-05

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this trail is to evaluate the performance of Genetron TERT/BRAF PCR Kit in Thyriod Cancer patients using real-time PCR method.

DETAILED DESCRIPTION:
This trial follows the principle of synchronous blinding. The enrolled cases are coded, and the enrolled samples are detected with Genetron TERT/BRAF PCR Kit and Sanger sequencing method. The results were determined independently according to the cutoff values or interpretation requirements provided by each method. The safety and effectiveness of this kit are confirmed and evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical diagnosis of suspected thyroid cancer who underwent fine-needle aspiration (FNA)
2. The sample should have corresponding basic clinical information, including: the patient's unique traceability number, age, gender, pathological diagnosis results, etc.
3. Subjects who can provide a complete FNA sample
4. Subjects who agree to provide follow-up diagnosis and treatment information

Exclusion Criteria:

1. The investigator considers that it is not appropriate to continue the clinical trial, such as the samples that are not prepared according to the required steps.
2. Samples with incomplete information required.
3. The amount of DNA extracted is not enough to complete the samples tested by the assessment reagent or comparative method.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital sample
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
The main purpose of this study is: by evaluating the Genetron TERT/BRAF PCR Kit to compare the results of the Sanger sequencing method, and to calculate the coincidence rate and consistency of the two methods. | 2 months

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Yunnan Cancer Hospital, Yunnan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT05395429/Prot_000.pdf